CLINICAL TRIAL: NCT00778063
Title: Intranasal Dexmedetomidine Decreases Emergence Delirium in Pediatric Patients After Sevoflurane Based General Anesthesia
Brief Title: Study Using Dexmedetomidine to Decreases Emergence Delirium in Pediatric Patients
Acronym: PED-DEX
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty enrolling patients
Sponsor: Ochsner Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2008.135.C
Record Dates: First submitted 2008-10-21; First posted 2008-10-23 (Estimated); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Otitis Media
Keywords: dexmedetomidine; pressure equalization tubes in the ear; myringotomy; sevoflurane
MeSH Terms: conditions — Otitis Media | interventions — Dexmedetomidine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- saline (Placebo Comparator): intranasal saline will be given 30 minutes prior to surgery
  Interventions: Drug: saline
- dexmedetomidine (Experimental): 2 mcg/kg dexmedetomidine will be given intranasally 30 minutes prior to surgery
  Interventions: Drug: dexmedetomidine

INTERVENTIONS:
Drug: dexmedetomidine — 2 mcg/kg intranasally 30 minutes prior to surgery
  Other Names: Precedex
  Arms: dexmedetomidine
Drug: saline — a volume of intranasal saline, calculated based on body weight, will be given 30 minutes prior to surgery
  Arms: saline

SUMMARY:
The purpose of this study is to evaluate the use of intranasal dexmedetomidine to reduce the incidence of emergence delirium during general sevoflurane anesthesia in a pediatric population receiving pressure equalization tubes in one or more ear.

DETAILED DESCRIPTION:
Emergence delirium has been described as a dissociated state of consciousness in which the child is irritable, uncompromising, uncooperative, incoherent, inconsolably crying, moaning, kicking or thrashing. The children can run the gambit from restlessness and incoherence to combative and psychotic. The incidence of emergence agitation or delirium is 80% after a procedure with sevoflurane-induced anesthesia.

Dexmedetomidine has been shown to have sedative and analgesic effects. In the pediatric population, it has been shown to provide sedation for radiographic procedures. Intravenously, it is has been shown to decrease emergence delirium following sevoflurane based anesthesia. The ability to administer a medication intranasally might solve the problem of emergence delirium and emergence agitation posed by the young patients undergoing myringotomy and tube placement.

ELIGIBILITY:
Inclusion Criteria:

* ASA class 1 or 2 (healthy patient or acute illness)
* Parental willingness to participate
* Candidate for pressure-equalization tubes (PET) as determined by the ENT department

Exclusion Criteria:

* ASA class 3 or 4 (chronic illness or life-threatening illness)
* Parental refusal to participate
* Significant liver disease by history
* Allergy to dexmedetomidine or midazolam
* Nasal deformity
* Fever in the three days prior to surgery
* Nausea or vomiting
* History of hypertension
* History of cardiac dysfunction/disorder
* Diabetes mellitus

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2008-09 (Actual); Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
To evaluate the use of intranasal dexmedetomidine to reduce the incidence of emergence delirium in general sevoflurane anesthesia. | 2 hours post-surgery

SECONDARY OUTCOMES:
Evaluate post-operative pain, emesis, and time to release from recovery. | 2 hours post-surgery

CONTACTS AND LOCATIONS:
Overall Officials: Usha Ramadhyani, MD, Principal Investigator — Ochsner Health System; Dominic S Carollo, MD, Study Director — Ochsner Health System
Locations (1):
- Ochsner Clinic Foundation, New Orleans, Louisiana, United States

REFERENCES:
- [Background] Olympio MA. Postanesthetic delirium: historical perspectives. J Clin Anesth. 1991 Jan-Feb;3(1):60-3. doi: 10.1016/0952-8180(91)90209-6. PMID 2007046
- [Result] Vlajkovic GP, Sindjelic RP. Emergence delirium in children: many questions, few answers. Anesth Analg. 2007 Jan;104(1):84-91. doi: 10.1213/01.ane.0000250914.91881.a8. PMID 17179249
- [Result] Cravero J, Surgenor S, Whalen K. Emergence agitation in paediatric patients after sevoflurane anaesthesia and no surgery: a comparison with halothane. Paediatr Anaesth. 2000;10(4):419-24. doi: 10.1046/j.1460-9592.2000.00560.x. PMID 10886700
- [Result] Mason KP, Zgleszewski SE, Dearden JL, Dumont RS, Pirich MA, Stark CD, D'Angelo P, Macpherson S, Fontaine PJ, Connor L, Zurakowski D. Dexmedetomidine for pediatric sedation for computed tomography imaging studies. Anesth Analg. 2006 Jul;103(1):57-62, table of contents. doi: 10.1213/01.ane.0000216293.16613.15. PMID 16790626
- [Result] Shukry M, Clyde MC, Kalarickal PL, Ramadhyani U. Does dexmedetomidine prevent emergence delirium in children after sevoflurane-based general anesthesia? Paediatr Anaesth. 2005 Dec;15(12):1098-104. doi: 10.1111/j.1460-9592.2005.01660.x. PMID 16324031
- [Result] Yuen VM, Irwin MG, Hui TW, Yuen MK, Lee LH. A double-blind, crossover assessment of the sedative and analgesic effects of intranasal dexmedetomidine. Anesth Analg. 2007 Aug;105(2):374-80. doi: 10.1213/01.ane.0000269488.06546.7c. PMID 17646493
- [Result] Yuen VM, Hui TW, Irwin MG, Yuen MK. A comparison of intranasal dexmedetomidine and oral midazolam for premedication in pediatric anesthesia: a double-blinded randomized controlled trial. Anesth Analg. 2008 Jun;106(6):1715-21. doi: 10.1213/ane.0b013e31816c8929. PMID 18499600
- [Result] Weldon BC, Bell M, Craddock T. The effect of caudal analgesia on emergence agitation in children after sevoflurane versus halothane anesthesia. Anesth Analg. 2004 Feb;98(2):321-326. doi: 10.1213/01.ANE.0000096004.96603.08. PMID 14742362
- [Result] Alhashemi JA, Daghistani MF. Effects of intraoperative i.v. acetaminophen vs i.m. meperidine on post-tonsillectomy pain in children. Br J Anaesth. 2006 Jun;96(6):790-5. doi: 10.1093/bja/ael084. Epub 2006 Apr 13. PMID 16613928
- [Result] Weldon BC, Watcha MF, White PF. Oral midazolam in children: effect of time and adjunctive therapy. Anesth Analg. 1992 Jul;75(1):51-5. doi: 10.1213/00000539-199207000-00010. PMID 1616162
- [Result] Guler G, Akin A, Tosun Z, Ors S, Esmaoglu A, Boyaci A. Single-dose dexmedetomidine reduces agitation and provides smooth extubation after pediatric adenotonsillectomy. Paediatr Anaesth. 2005 Sep;15(9):762-6. doi: 10.1111/j.1460-9592.2004.01541.x. PMID 16101707
- [Result] Meistelman C, Plaud B, Donati F. Rocuronium (ORG 9426) neuromuscular blockade at the adductor muscles of the larynx and adductor pollicis in humans. Can J Anaesth. 1992 Sep;39(7):665-9. doi: 10.1007/BF03008227. PMID 1394754